CLINICAL TRIAL: NCT00898027
Title: Pilot Study of the Effects of Epidermal Growth Factor Receptor (EGFR) Inhibitors on Magnesium Homeostasis
Brief Title: Effect of Epidermal Growth Factor Receptor Inhibitors on Magnesium Homeostasis in Patients With Cancer
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Laura W. Goff, MD, Assistant Professor of Medicine; Associate Director, Hematology/Oncology, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0615; VU-VICC-GI-0615; VU-VICC-IRB-060364
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: laboratory biomarker analysis — laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and urine in the laboratory from patients with cancer receiving epidermal growth factor receptor inhibitors may help doctors understand the effect of epidermal growth factor receptor inhibitors on magnesium levels in the body.

PURPOSE: This laboratory study is looking at the effect of epidermal growth factor receptor inhibitors on magnesium homeostasis in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of EGFR inhibitors on magnesium homeostasis in patients with cancer.

OUTLINE: This is a pilot study.

Patients undergo blood and urine sample collection at baseline and at 2, 4, and 8 weeks during treatment.

After finishing treatment, patients are followed periodically for up to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of malignancy

  * Planning to receive therapy with an inhibitor of the EGFR pathway (either on or off a clinical trial and may be monotherapy or combined with other therapies)
* Normal serum magnesium level

Exclusion Criteria:

* Glomerular filtration rate ≥ 60 mL/min
* No severe underlying renal dysfunction
* Normal serum potassium and calcium level
* No history of primary or secondary hyperparathyroidism

PRIOR CONCURRENT THERAPY:

* No prior EGFR pathway inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with the diagnosis of a malignancy for which they are considering therapy with an inhibitor of the EGFR pathway, have received an inhibitor of the EGFR pathway prior to study start, have no severe underlying renal dysfunction as defined as estimated GFR<60 by MDRD equation and must be ≥ 18 years of age.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Effects of EGFR inhibitors on magnesium homeostasis | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goff, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center